CLINICAL TRIAL: NCT04965857
Title: Comparison of the Hologic Genius Digital Diagnostics System With the Liquid-based Cytology (LBC) Manual Microscopic Approach
Brief Title: Comparison of the Hologic Genius Digital Diagnostics System With the Liquid-based Cytology (LBC) Manual Microscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hologic Deutschland GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: BTS1650_20
Record Dates: First submitted 2021-06-16; First posted 2021-07-16 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Cervical Cancer Screening

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Slides from the German Co-Screening program: From 25,000 LBC slides (ThisPrep, Hologic Inc., USA) from the German Co-screening program evaluated using the Genius Digital cytology system all abnormal findings according to Munich III groups (II-p - V) and each 10th normal slide (Munich III group I and II) will be selected for the prospective evaluation by manual microscopy.
  Interventions: Diagnostic Test: Hologic's Genius Digital Diagnostics System

INTERVENTIONS:
Diagnostic Test: Hologic's Genius Digital Diagnostics System — Genius Digital Diagnostics is a digital cytology platform to combine a new artificial intelligence (AI) algorithm with advanced volumetric imaging technology to help cytotechnologists and pathologists identify pre-cancerous lesions and cancer cells in women.

SUMMARY:
Quality assurance of the laboratory examinations. Prospective non-interventional study with ThinPrep slides collected during the German Co-Screening Program and routinely sent to the lab to prospectively evaluate the clinical performance of the Hologic Genius Digital Cytology (DC) system vs. the liquid-based cytology (LBC) manual microscopic approach

DETAILED DESCRIPTION:
The cause of cervical cancer is a persistent infection with high-risk types of human papillomavirus (HPV). Cytology has been the gold standard for cervical screening since the introduction of routine screening with the Pap test in the 1950s due to its effect on mortality in regions with screening programs. Since that time, there have been several technological advances (LBC, Imaging) to improve and automate cervical cytology, resulting in increased disease detection and efficiency. The Hologic's Genius Digital Diagnostics System is a CE-IVD (CE-marked in vitro diagnostic device) marked digital cytology platform. For quality assurance and to prospectively evaluate the Hologic Genius Digital Cytology (DC) system in the lab, selected routinely screened and already archived slides will be additionally reviewed with the liquid-based cytology (LBC) manual microscopic approach. Only anonymized results will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* LBC ThinPrep® samples are collected by gynaecologists and sent routinely to cytology laboratory Zotz & Klimas as part of the German Cervical cancer screening program.

Ages: 35 Years to 90 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: As part of the German National Cancer Plan, women over the age of 35 years will be given a co-test comprising a Pap smear and an HPV test, every three years.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of detection of pre-cancerous lesions using Hologic Genius Digital Cytology Imaging scanner. | 1 year
  To demonstrate non-inferiority, the appropriate approximative one-sided 95% confidence interval for the true difference between the two approaches (Digital Cytology and Manual microscopic reading) will be constructed.

SECONDARY OUTCOMES:
To assess the rate of inadequate slides that cannot be read by the Hologic Genius Digital Cytology system. | 1 year
Change in time needed to screen 80 slides using Hologic Genius Digital Cytology Imaging scanner. | 1 year
  To assess the impact on the workflow of the introduction of a Digital Cytology procedure to a high-throughput screening lab in Germany.
Clinical performance of Hologic Genius Digital Cytology Imaging scanner using cells on a ThinPrep® slide. | 1 year
  The performance of Hologic Genius Digital Cytology Imaging scanner during cervical cancer screening (using histology as reference method) will be assessed via sensitivity, specificity, positive and negative predictive values.

CONTACTS AND LOCATIONS:
Locations (1):
- Zotz Klimas Partner für Diagnostik und Prävention MVZ Düsseldorf-Centrum, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No